CLINICAL TRIAL: NCT00615784
Title: A Phase II Study of Bexarotene in Patients With Acute Myeloid Leukemia
Brief Title: Phase II Study of Bexarotene in Patients With Acute Myeloid Leukemia
Acronym: UPCC04407
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated. Eisai's Targretin acquired by another pharmaceutical company.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04407; UPCC 04407
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; Bexarotene
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Bexarotene

INTERVENTIONS:
Drug: Bexarotene — Bexarotene given orally at a dose of 300mg/m2 until disease progression or unacceptable toxicities experienced by patient

SUMMARY:
The purpose of this study is to evaluate the activity of bexarotene, a retinoic acid class drug, in patients with Acute Myeloid Leukemia (AML) that has returned after or is resistant to standard chemotherapy or are otherwise not eligible for conventional chemotherapy. Retinoic acids are a class of drugs related to Vitamin A, and have a wide range of effects within normal and malignant cells that affect cell growth and cell death.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Confirmed diagnosis of AML as proven by bone marrow biopsy
* Must have received prior induction therapy with conventional chemotherapy and/or Mylotarg or otherwise not eligible for conventional chemotherapy
* ECOG performance status of 0-2
* Recovered from toxicities of prior chemotherapy

Exclusion Criteria:

* History of pancreatitis
* Active alcohol abuse
* Taken bexarotene in the past
* WBC > 10,000/uL at time of enrollment
* Cytotoxic therapy within the past 14 days other than hydrea, low dose cytarabine or low dose Mylotarg
* Significant organ disfunction: total bilirubin > 3x ULN, AST or ALT >3 x ULN, creatinine > 3 mg/dL, on blood pressure supporting medications or mechanical ventilation
* Active participant in any other investigational treatment study for AML
* Life expectancy of less than 1 month
* Use of blood growth factors (G-CSF, GM-CSF, Aranesp, erythropoietin, or Neumega) within 1 week prior to treatment initiation
* Uncontrolled hyperlipidemia
* Known history of HIV
* Known active CNS involvement with AML
* Women of childbearing potential or active breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05-25 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2013-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald E. Tsai, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bexarotene 300mg/m2 Daily: Bexarotene: Bexarotene given orally at a dose of 300mg/m2 until disease progression or unacceptable toxicities experienced by patient
Period: Overall Study
Arm/Group | Bexarotene 300mg/m2 Daily
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This study was completed several years ago, and the principal investigator has left the institution. Limited records are available, and despite our best efforts data are only available for 14 of the 24 enrolled participants.
Groups:
- Bexarotene 300mg/m2: Bexarotene: Bexarotene given orally at a dose of 300mg/m2 until disease progression or unacceptable toxicities experienced by patient
Arm/Group | Bexarotene 300mg/m2
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 74 [20 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response Rate of Bexarotene Monotherapy in Subjects With Relapsed/Refractory AML or Newly Diagnosed AML Who Are Unable to Receive Systemic Chemotherapy.
Description: Hematologic response will be assessed according to modified criteria of an international working group defined by Cheson et al, Report of an international working group to standardize response criteria for myelodysplastic syndromes. Blood, 1 December 2000, Vol. 96, No. 12, pp. 3671-3674
Time Frame: Two months after 17th patient has started treatment with Bexarotene, for up to 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Bexarotene 300mg/m2
Number analyzed (Participants) | 14
Participants | 1

2. Secondary Outcome: Bone Marrow Response Rate of Bexarotene in Subjects With AML Unable/Unwilling to Receive Systemic Chemotherapy
Description: A clinically significant result will be recorded if the patient's bone marrow blasts percentage decreased by 50% or more over pretreatment blast percentage.
Time Frame: Two months after 17th patient has started treatment with Bexarotene, up to 1 year.
Population: This study was completed several years ago, and the principal investigator has left the institution. Limited records are available, and despite our best efforts data are only available for 14 of the 24 enrolled participants. Additionally only 5 patients had a bone marrow biopsy at 2 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Bexarotene 300mg/m2
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Arm/Group | Bexarotene 300mg/m2
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexarotene 300mg/m2 (N=14)
hypothyroidism (Endocrine disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes